CLINICAL TRIAL: NCT05933070
Title: A Phase I Open-Label Dose Escalation Study Of Intravenous INKmune In Patients With Myelodysplastic Syndrome With Excess Blasts (MDS-EB-1/2 - MDS-CMML 1/2) Or Acute Myeloid Leukaemia (AML)
Brief Title: A Phase I Open-Label Dose Escalation Study of Intravenous INKmune In Patients With MDS or AML
Acronym: LAUREL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow/low Enrollment
Sponsor: Inmune Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INMB-INB16-002
Record Dates: First submitted 2023-06-02; First posted 2023-07-06 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Cancer; MDS-EB; Myelodysplastic Syndromes; Acute Myeloid Leukemia; AML
Keywords: MDS; AML; NK Cell Based Therapy; Immune Based Therapy
MeSH Terms: conditions — Neoplasms; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Participants will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15 in addition to supportive care. Three cohorts, comprised of at least 3 participants, are planned. Each participant will be screened up to 28 days prior to treatment. After participants have received all doses, they will be reviewed at Day 29 and Day 43 and then followed up with monthly clinic appointments for the following 3 months (Days 73 and 119) for clinical assessment and blood tests. Once Day 119 visit is completed this classifies end of study for the participant. The trial will end after data collection has been completed for each trial participant.
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schedule of Assessments (Experimental): INKmune therapy will be administered by a slow intravenous injection via conventional blood giving set. Patients will receive 3 weekly IV doses of INKmune on Day 1, 8, and 15.
  * In Cohort 1, the initial planned dose is 1 x 10^8 INKmune;
  * In Cohort 2, the weekly dose will increase to 3 x 10^8 INKmune;
  * In Cohort 3, the weekly dose will increase to 5 x 10^8 INKmune.
  Interventions: Biological: INKmune

INTERVENTIONS:
Biological: INKmune — INKmune is a patented biologic delivery system and method for cancer treatment using in vivo priming and activation of natural killer (NK) cells in order to achieve tumor cell lysis. INKmune is a suspension of INB16 cells which have been rendered replication incompetent. INKumne is a replication-incompetent tumor cell line that does not require donor matching.

SUMMARY:
INMB-INB16-002 is a Phase I open-label, dose escalation study of INKmune therapy in subjects with myelodysplastic syndrome (MDS) with excess blasts without Auer rods (EB-1 or 2, or CMML 1 or 2) or subjects with acute myeloid leukaemia (AML) in complete remission.

DETAILED DESCRIPTION:
INMB-INB16-002 is a Phase 1 open-label, dose escalation study of INKmune therapy in subjects with MDS with excess blasts without Auer rods (EB-1 or 2, or CMML 1 or 2) who have completed treatment with Azacytidine (AZA) and not achieved complete remission (CR) and who are not thought to be fit for intensive chemotherapy, or subjects with AML in complete remission (or complete remission with incomplete count recovery) unsuitable for intensive chemotherapy or allogeneic stem cell transplantation or subjects with relapsed MDS or AML post-allogeneic stem cell transplant with slowly progressive disease unsuitable for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subjects with:

   1. MDS-EB-1/2, MDS-CMML 1-2 who have completed treatment with Azacytidine (AZA), and not achieved complete remission (CR) who are not thought to be fit for intensive chemotherapy.
   2. Subjects with AML in complete remission (or complete remission with incomplete count recovery) unsuitable for intensive chemotherapy or allogeneic stem cell transplantation.
   3. Subjects with relapsed MDS or AML post-allogeneic stem cell transplant, with slowly progressive disease unsuitable for intensive chemotherapy.
3. Subject has adequate organ and marrow function (as defined below):

   1. Serum creatinine ≤ 1.5 X ULN, or measured creatinine clearance ≥ 60 ml/min/1.73m2.
   2. Aspartate aminotransferase (AST) and ALT levels ≤ 3 X ULN.
   3. Total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome.
   4. Absolute neutrophil (ANC) ≥ 500/mm3; 0.5 x 109/L
   5. Platelet count ≥ 50,000/mm3; 50 x 109/L
   6. Haemoglobin ≥ 100mg/L (transfusion to obtain haemoglobin ≥ 100mg/L within 24 hours prior to dosing is allowed).
4. Subject must be at least 21 days from previous anticancer therapy (eg, chemotherapy, radiation therapy, immunotherapy and monoclonal antibodies, or investigational therapeutic agents) at the time of study screening and meet criteria in "3" above.
5. Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. a. Sexually active female subjects of childbearing potential must agree to use a highly effective method of contraception for the duration of study therapy and for 3 months after the last dose of INKmune. Acceptable forms of contraception methods are as follows:

   * Non-hormonal methods (i.e. intrauterine device, IUD)
   * have vasectomised partner (the vasectomised partner must be the sole partner of the trial participant and have received medical assessment of its surgical success)
   * True sexual abstinence Women of childbearing potential must discontinue any hormonal forms of birth control at least 4 weeks prior to first study dosing and commence using a highly effective, non- hormonal method as described above. Any pregnancy that occurs for study participants should be monitored for potential side effects.

     b. Male subjects with partners who are of childbearing potential must agree a double barrier method of contraception i.e. condom with either cap or diaphragm for the duration of study therapy and for 3 months after the last dose of INKmune. Male subjects with partners who are pregnant must use a condom for the same duration to avoid INKmune exposure to developing foetus. Note: Subjects who are abstinent (defined as refraining from heterosexual intercourse during the entire period of risk associated with study treatments), must agree to remain abstinent for the study duration and for 3 months after the last study dose of INKmune. The reliability of sexual abstinence will be evaluated in relation to the preferred and usual lifestyle of the subject.
7. Subject, must be able to understand and voluntarily sign a written informed consent, and are willing and able to comply with the protocol requirements.
8. Subject must have a life expectancy greater than 3 months in the opinion of the PI.

Exclusion Criteria:

1. Subject diagnosed with any other sub-classification of MDS.
2. Subject is currently receiving cancer-specific treatment with the exceptions of supportive treatments such as bisphosphonate or steroid treatments for symptomatic control.
3. Subject has had prior NK cell targeting therapy.
4. Subject has a current requirement for steroids > 10 mg daily; prednisolone or equivalent.
5. Subject has impaired cardiac function or clinically significant cardiac disease including the following:

   1. New York Heart Association grade III or IV congestive heart failure.
   2. Myocardial infarction within the last 6 months prior to dosing with INKmune
   3. Impaired left ventricular ejection fraction (LVEF < 40%) as assessed according to institutional standards.
6. Subject has shown lack of recovery of prior AEs to Grade ≤1 severity (NCI CTCAE v5.0) (except alopecia) due to therapy administered prior to the initiation of study drug dosing. Stable persistent grade 2 peripheral neuropathy may be allowed as determined on a case-by-case basis at the discretion of the PI and Medical Monitor.
7. Subject has known allergy to any of the formulation components of INKmune.
8. Subjects has active, severe infection requiring systemic treatment. Subjects may become eligible once infection has resolved and they are at least seven days from completion of antibiotics.
9. Subject concomitant use of complementary or alternative medication or other agents (investigational therapeutic agents) will not be allowed without approval of a PI or sub- investigator (SI). Every effort will be made to maximize subject safety and minimize changes in chronic medications.
10. Subject is pregnant or is currently breastfeeding.
11. Subject has uncontrolled seizures as determined by the PI.
12. Subject has any other condition or finding that in the opinion of the PI or Sponsor Medical Monitor may render the subject at excessive risk for treatment complications or may not be able provide evaluable outcome information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Primary Objective 1 | 2-3 years
  Identify the incidence and seriousness of AEs and their relationship (causality) to INKmune as graded by NCI CTCAE criteria v.5.0.
Primary Objective 2 | 2-3 years
  Identify a RP2D of INKmune. The RP2D is defined as the maximum tolerated dose (MTD) of the agent which will be defined as the dose at which the complication rate is less than 33%.

SECONDARY OUTCOMES:
Secondary Objective 1 | 1-2 years
  To assess the overall response rate by measuring changes in percentage blasts in PB at days 29, 43, 73, 119 and BM at day 29.
Secondary Objective 2 | 3-4 years
  To assess the overall response rate, partial response rate or complete response rate in subjects administered INKmune using the WHO criteria by measuring changes in vital signs, electrocardiogram (ECG), and safety laboratory parameters throughout the study.
Secondary Objective 3 | 2-3 years
  To assess the progression-free survival (PFS) time defined as time to increase in transfusion dependence and or increase in percentage blasts in Peripheral Blood (PB) and/or Bone Marrow (BM).

OTHER OUTCOMES:
Exploratory Objective 1 | 2-3 years
  Assess the pharmacodynamics (PD) (proof of biology) of INKmune by analyzing NK cells obtained from peripheral blood, and bone marrow as available and to measure primed NK cells and cell kill ability using the tumour killing assay.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Kay-Mindick, Study Director — INmune Bio
Locations (3):
- Attikon University General Hospital, Athens, Attica, Greece
- United Kingdom (2):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Sheffield Teaching Hospitals NHS FT - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arai S, Meagher R, Swearingen M, Myint H, Rich E, Martinson J, Klingemann H. Infusion of the allogeneic cell line NK-92 in patients with advanced renal cell cancer or melanoma: a phase I trial. Cytotherapy. 2008;10(6):625-32. doi: 10.1080/14653240802301872. PMID 18836917
- [Background] Bengala, C., V. Rasini, R. Sternieri, M. Dominici, A. Andreotti, R. Gelmini, L. Cafarelli, P. Bevini, A. Berti, and P. Conte. 2007. 'Phase I study of intraperitoneal MHC unrestricted adoptive cell therapy with TALL-104 cells in patients with peritoneal carcinosis', Journal of Clinical Oncology, 25: 3054-54.
- [Background] Bryceson YT, March ME, Ljunggren HG, Long EO. Activation, coactivation, and costimulation of resting human natural killer cells. Immunol Rev. 2006 Dec;214:73-91. doi: 10.1111/j.1600-065X.2006.00457.x. PMID 17100877
- [Background] Carlsten M, Baumann BC, Simonsson M, Jadersten M, Forsblom AM, Hammarstedt C, Bryceson YT, Ljunggren HG, Hellstrom-Lindberg E, Malmberg KJ. Reduced DNAM-1 expression on bone marrow NK cells associated with impaired killing of CD34+ blasts in myelodysplastic syndrome. Leukemia. 2010 Sep;24(9):1607-16. doi: 10.1038/leu.2010.149. Epub 2010 Jul 8. PMID 20613786
- [Background] Carlsten M, Norell H, Bryceson YT, Poschke I, Schedvins K, Ljunggren HG, Kiessling R, Malmberg KJ. Primary human tumor cells expressing CD155 impair tumor targeting by down-regulating DNAM-1 on NK cells. J Immunol. 2009 Oct 15;183(8):4921-30. doi: 10.4049/jimmunol.0901226. PMID 19801517
- [Background] Cesano A, Santoli D. Two unique human leukemic T-cell lines endowed with a stable cytotoxic function and a different spectrum of target reactivity analysis and modulation of their lytic mechanisms. In Vitro Cell Dev Biol. 1992 Sep-Oct;28A(9-10):648-56. doi: 10.1007/BF02631041. PMID 1429367
- [Background] Chandhok NS, Boddu PC, Gore SD, Prebet T. What are the most promising new agents in myelodysplastic syndromes? Curr Opin Hematol. 2019 Mar;26(2):77-87. doi: 10.1097/MOH.0000000000000483. PMID 30632987
- [Background] Epling-Burnette PK, Bai F, Painter JS, Rollison DE, Salih HR, Krusch M, Zou J, Ku E, Zhong B, Boulware D, Moscinski L, Wei S, Djeu JY, List AF. Reduced natural killer (NK) function associated with high-risk myelodysplastic syndrome (MDS) and reduced expression of activating NK receptors. Blood. 2007 Jun 1;109(11):4816-24. doi: 10.1182/blood-2006-07-035519. Epub 2007 Mar 6. PMID 17341666
- [Background] Fehniger TA, Miller JS, Stuart RK, Cooley S, Salhotra A, Curtsinger J, Westervelt P, DiPersio JF, Hillman TM, Silver N, Szarek M, Gorelik L, Lowdell MW, Rowinsky E. A Phase 1 Trial of CNDO-109-Activated Natural Killer Cells in Patients with High-Risk Acute Myeloid Leukemia. Biol Blood Marrow Transplant. 2018 Aug;24(8):1581-1589. doi: 10.1016/j.bbmt.2018.03.019. Epub 2018 Mar 27. PMID 29597002
- [Background] Fozza C. The burden of autoimmunity in myelodysplastic syndromes. Hematol Oncol. 2018 Feb;36(1):15-23. doi: 10.1002/hon.2423. Epub 2017 Apr 27. PMID 28449370
- [Background] Gong JH, Maki G, Klingemann HG. Characterization of a human cell line (NK-92) with phenotypical and functional characteristics of activated natural killer cells. Leukemia. 1994 Apr;8(4):652-8. PMID 8152260
- [Background] Hou HA, Tsai CH, Lin CC, Chou WC, Kuo YY, Liu CY, Tseng MH, Peng YL, Liu MC, Liu CW, Liao XW, Lin LI, Yao M, Tang JL, Tien HF. Incorporation of mutations in five genes in the revised International Prognostic Scoring System can improve risk stratification in the patients with myelodysplastic syndrome. Blood Cancer J. 2018 Apr 4;8(4):39. doi: 10.1038/s41408-018-0074-7. PMID 29618722
- [Background] Kiladjian JJ, Bourgeois E, Lobe I, Braun T, Visentin G, Bourhis JH, Fenaux P, Chouaib S, Caignard A. Cytolytic function and survival of natural killer cells are severely altered in myelodysplastic syndromes. Leukemia. 2006 Mar;20(3):463-70. doi: 10.1038/sj.leu.2404080. PMID 16408099
- [Background] Kottaridis PD, North J, Tsirogianni M, Marden C, Samuel ER, Jide-Banwo S, Grace S, Lowdell MW. Two-Stage Priming of Allogeneic Natural Killer Cells for the Treatment of Patients with Acute Myeloid Leukemia: A Phase I Trial. PLoS One. 2015 Jun 10;10(6):e0123416. doi: 10.1371/journal.pone.0123416. eCollection 2015. PMID 26062124
- [Background] Lanier LL. Up on the tightrope: natural killer cell activation and inhibition. Nat Immunol. 2008 May;9(5):495-502. doi: 10.1038/ni1581. PMID 18425106
- [Background] Loghavi S, Sui D, Wei P, Garcia-Manero G, Pierce S, Routbort MJ, Jabbour EJ, Pemmaraju N, Kanagal-Shamanna R, Gur HD, Hu S, Zuo Z, Medeiros LJ, Kantarjian HM, Khoury JD. Validation of the 2017 revision of the WHO chronic myelomonocytic leukemia categories. Blood Adv. 2018 Aug 14;2(15):1807-1816. doi: 10.1182/bloodadvances.2018019224. PMID 30054307
- [Background] Lucas M, Schachterle W, Oberle K, Aichele P, Diefenbach A. Dendritic cells prime natural killer cells by trans-presenting interleukin 15. Immunity. 2007 Apr;26(4):503-17. doi: 10.1016/j.immuni.2007.03.006. Epub 2007 Mar 29. PMID 17398124
- [Background] Nazha A, Bejar R. Molecular Data and the IPSS-R: How Mutational Burden Can Affect Prognostication in MDS. Curr Hematol Malig Rep. 2017 Oct;12(5):461-467. doi: 10.1007/s11899-017-0407-9. PMID 28844082
- [Background] North J, Bakhsh I, Marden C, Pittman H, Addison E, Navarrete C, Anderson R, Lowdell MW. Tumor-primed human natural killer cells lyse NK-resistant tumor targets: evidence of a two-stage process in resting NK cell activation. J Immunol. 2007 Jan 1;178(1):85-94. doi: 10.4049/jimmunol.178.1.85. PMID 17182543
- [Background] Papaemmanuil E, Gerstung M, Malcovati L, Tauro S, Gundem G, Van Loo P, Yoon CJ, Ellis P, Wedge DC, Pellagatti A, Shlien A, Groves MJ, Forbes SA, Raine K, Hinton J, Mudie LJ, McLaren S, Hardy C, Latimer C, Della Porta MG, O'Meara S, Ambaglio I, Galli A, Butler AP, Walldin G, Teague JW, Quek L, Sternberg A, Gambacorti-Passerini C, Cross NC, Green AR, Boultwood J, Vyas P, Hellstrom-Lindberg E, Bowen D, Cazzola M, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Clinical and biological implications of driver mutations in myelodysplastic syndromes. Blood. 2013 Nov 21;122(22):3616-27; quiz 3699. doi: 10.1182/blood-2013-08-518886. Epub 2013 Sep 12. PMID 24030381
- [Background] Sabry M, Lowdell MW. Tumor-primed NK cells: waiting for the green light. Front Immunol. 2013 Nov 25;4:408. doi: 10.3389/fimmu.2013.00408. PMID 24324471
- [Background] Sabry M, Zubiak A, Hood SP, Simmonds P, Arellano-Ballestero H, Cournoyer E, Mashar M, Pockley AG, Lowdell MW. Tumor- and cytokine-primed human natural killer cells exhibit distinct phenotypic and transcriptional signatures. PLoS One. 2019 Jun 26;14(6):e0218674. doi: 10.1371/journal.pone.0218674. eCollection 2019. PMID 31242243
- [Background] Tsirogianni M, Grigoriou E, Kapsimalli V, Dagla K, Stamouli M, Gkirkas K, Konsta E, Karagiannidou A, Gkodopoulos K, Stavroulaki G, Pappa V, Angelopoulou M, Lowdell M, Tsirigotis P. Natural killer cell cytotoxicity is a predictor of outcome for patients with high risk myelodysplastic syndrome and oligoblastic acute myeloid leukemia treated with azacytidine. Leuk Lymphoma. 2019 Oct;60(10):2457-2463. doi: 10.1080/10428194.2019.1581935. Epub 2019 Apr 5. PMID 30947589
- [Background] Tonn T, Schwabe D, Klingemann HG, Becker S, Esser R, Koehl U, Suttorp M, Seifried E, Ottmann OG, Bug G. Treatment of patients with advanced cancer with the natural killer cell line NK-92. Cytotherapy. 2013 Dec;15(12):1563-70. doi: 10.1016/j.jcyt.2013.06.017. Epub 2013 Oct 1. PMID 24094496
- [Background] Visonneau S, Cesano A, Porter DL, Luger SL, Schuchter L, Kamoun M, Torosian MH, Duffy K, Sickles C, Stadtmauer EA, Santoli D. Phase I trial of TALL-104 cells in patients with refractory metastatic breast cancer. Clin Cancer Res. 2000 May;6(5):1744-54. PMID 10815893
- [Background] Williams BA, Law AD, Routy B, denHollander N, Gupta V, Wang XH, Chaboureau A, Viswanathan S, Keating A. A phase I trial of NK-92 cells for refractory hematological malignancies relapsing after autologous hematopoietic cell transplantation shows safety and evidence of efficacy. Oncotarget. 2017 Jul 12;8(51):89256-89268. doi: 10.18632/oncotarget.19204. eCollection 2017 Oct 24. PMID 29179517